CLINICAL TRIAL: NCT02147704
Title: Effect of High- and Low-sodium Intake on the Pharmacokinetics and Pharmacodynamic Effects of Fimasartan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DongGuk University (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Moo-Yong Rhee, Professor, MD, PhD, Director of Clinical Trial Center, DongGuk University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DUMC-FMS-NA
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goup I (Other): Group I: Fimasartan 60 mg in a low-sodium intake period --> Fimasartan 60 mg in a high-sodium intake period
  Interventions: Dietary Supplement: High-sodium diet; Dietary Supplement: low-sodium diet
- Group II (Other): Group II: Fimasartan 60 mg in a high-sodium intake period --> Fimasartan 60 mg in a low-sodium intake period
  Interventions: Dietary Supplement: High-sodium diet; Dietary Supplement: low-sodium diet

INTERVENTIONS:
Dietary Supplement: High-sodium diet — 1. One of high- or low sodium intake for 7 days during each period
  2. High sodium intake: 50 mmol/day by diet + 250 mmol/day by salt tablets
Dietary Supplement: low-sodium diet — 1. One of high- or low sodium intake for 7 days during each period
  2. Low sodium intake : 50 mmol/day by diet

SUMMARY:
It has been known that the blood pressure lowering effect of angiotensin receptor antagonists (ARBs) and angiotensin converting enzyme (ACE) inhibitors is impaired in patients on high sodium intake. There was an enhanced blood pressure lowering effect of ACE inhibitor when sodium intake was restricted or diuretics were added.

The reason is partially explained by sodium sensitivity or low rennin activity in high sodium intake. However, the exact mechanism of sodium intake dependency is not clearly understood.

In a recent study, an ARB, candesartan was revealed to have sodium intake dependency, showing lower plasma concentration when subjects were on high sodium intake compared to on low sodium intake. However, plasma concentration of another ARB, valsartan and an ACE inhibitor ramipril was not changed depending on the sodium intake.

The strongly suggested mechanism is the involvement of transporter P-glycoprotein (Pg-P). the function and expression of Pg-P are modified by genetic polymorphism of multidrug resistance 1 gene.

Although the transport mechanism of Fimasartan from gut is not fully understood, it has been known that the multidrug resistance 1 is not involved. Thus, the pharmacokinetic and pharmacodynamic property of fimasartan is expected not to be affected by the status of sodium intake.

The present study is designed to investigate whether the pharmacokinetic and pharmacodynamic property of fimasartan is changed depending on the sodium intake.

DETAILED DESCRIPTION:
The study design is a two-diet, two-period, two-sequence, randomized, open label and cross-over with 1-week diet-washout and 2-weeks drug-washout interval. The participants (n=16) are randomly assigned to either of 7 days of low sodium (50 mmol/day) or high sodium diet (300 mol) after hospitalization. After completion of 7-days of first period, all participants are discharge and recommended to eat usual diet. After 1-week of diet washout, all participants are hospitalized for second period. The compliance of diet is determined by measurement of 24-hour urine sodium excretion. The 24-hour urine sodium excretion should be < 100 mmol/24-hour in the low sodium diet period and > 200 mmol/24-hour in high sodium diet period.

On the morning of 7th day of each period (high sodium or low sodium diet period), all participants receive 60 mg of fimasartan in the fasting state. Blood samples for pharmacokinetic and pharmacodynamic study are drawn for 24-hour.

The detailed measures are as followings:

1. High- and low-sodium intake

   1. One of high- or low sodium intake for 7 days during each period
   2. Low sodium intake : 50 mmol/day by diet
   3. High sodium intake: 50 mmol/day by diet + 250 mmol/day by salt tablets
2. 24 hour excreted amount of sodium in urine to determine the compliance for the high- and low-sodium intake

   1. 24 hour excreted amount of sodium in urine for low sodium intake < 100 mmol
   2. 24 hour excreted amount of sodium in urine for high sodium intake > 200 mmol
3. Vital signs

   a. Systolic and diastolic blood pressures and pulse rate in sitting position and body temperature
4. Blood chemistry and complete blood count

   1. Measure at the morning of first day after overnight fasting
   2. white blood cell count, red blood count, hemoglobin, hematocrit, platelet, Calcium, sodium, potassium, glucose, blood urea nitrogen, creatinine, uric acid, cholesterol, albumin, total bilirubin, AST, ALT, blood urea nitrogen
5. Urinalysis

   a. potential of hydrogen, protein, bilirubin, glucose, urobilinogen, ketone, nitrite, blood
6. Pharmacokinetic blood sampling

   a. Plasma samples for fimasartan concentration
7. Pharmacodynamic blood sampling

   1. Plasma samples for renin activity
   2. Serum samples for aldosterone concentration

ELIGIBILITY:
Inclusion Criteria:

* The subject who has a body weight of 50 to 90 kg and has a body mass index (BMI) of 18.5 to 29.9 kg/m2.
* The subject who voluntarily agrees to participate in the study by written informed consent.

Exclusion Criteria:

* The subject who has a history of hypersensitivity reaction to fimasartan or other drugs.
* The subject who has galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* The subject who has a history of any history or evidence of any clinically significant hepatic, urologic, gastrointestinal, neurologic, pulmonary, endocrinologic, musculoskeletal, hematologic, oncologic, psychiatric, cardiovascular disease.
* The subject who has a history of gastrointestinal disease (Crohn's disease, ulcer, acute or chronic pancreatitis and etc.) or surgery (except simple appendectomy or hernia repair) which can significantly affect the absorption of the study drug.
* The subject who has a systolic blood pressure (SBP) =<90 or >=160 mmHg, diastolic blood pressure (DBP) =<60 or >=90 mmHg, and/or pulse rate (PR) >=100.
* The subject who has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 x upper limit of normal.
* The subject who has a history of drug abuse.
* The subject who has participated in any interventional clinical study within 60 days prior to the study drug administration.
* The subject who has used any prescribed or traditional oriental drugs within 2 weeks, or nonprescribed drugs within 1 week prior to the study administration.
* The subject who has donated 1 unit (450 mL) of blood or more within 60 days, or received a transfusion of any blood or blood products or donated plasma within 60 days prior to the study administration.
* The subject who has eaten unusual diet which can affect the absorption, distribution, metabolism, elimination processes of the study drug.
* The subject who is a heavy smoker (>10 cigarettes per day) within 3 months prior to Screening and unable to quit smoking during study period.
* The subject who consumes more than 21 unit/week of alcohols or unable to stop drinking during study period.
* The subjects who consumes excessive amount of grapefruit containing beverage of food and unable to quit eating or drinking them.
* The subjects who consumes excessive amount of caffeine containing beverage of food and unable to quit eating or drinking them.
* The subject who has a positive result for hepatitis C antibodies, hepatitis B surface antigen,
* The subject who are unable to perform the present clinical study, judged by investigators.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time 0 to 24 hr (AUC0-24h) and area under the curve form time 0 to infinite (AUC0-inf) of the study drug in each diet period | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr after dose

SECONDARY OUTCOMES:
Cmax of the study drug in each diet period | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr after dose

OTHER OUTCOMES:
Change of plasma renin activity and plasma aldosterone level from the baseline in each diet period | -24, -22, -20, -18, -16, and -12 hr before dose and predose, 2, 4, 6, 8, 12, and 24 h after dose
Tmax and half-life of the study drug in each diet period | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr after dose

CONTACTS AND LOCATIONS:
Overall Officials: Moo-Yong Rhee, MD, PhD, Principal Investigator — Clinical Trial Center, Dongguk University Ilsan Hospital
Locations (1):
- Clinical Trial Center, Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea